CLINICAL TRIAL: NCT00185757
Title: Cytokine Induced Killer Cells as Post-Transplant Immunotherapy Following Allogeneic Hematopoietic Cell Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Robert Negrin (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Robert Negrin, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT162; 95070; BMT162; NCT00185757; 13644 (Other: Stanford IRB)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Multiple Myeloma; Blood and Marrow Transplant (BMT)
MeSH Terms: conditions — Multiple Myeloma

ARMS (1):
- Cytokine-induced Killer Cells (Experimental): The first cohort =1X10 7 cf expanded cells/kg. The second cohort = 5x10 7 expanded cells/kg. The second cohort = 1X10 8 expanded cells/kg.
  Interventions: Drug: Cytokine Induced Killer Cells

INTERVENTIONS:
Drug: Cytokine Induced Killer Cells — CIK cell dose escalation will be performed in cohorts of three patients per group. The initial dose utilized will be 1x107 expanded cells/kg. Previously, unmanipulated donor lymphocytes administered at this dose did not result in significant GVHD 7. The expansion of the CIK cell population is expected to diminish the T cell subsets responsible for GVHD further reducing the risk of GVHD to recipients. The dose will be increased to 5x107 expanded cells/kg and 1x108 expanded cells/kg in successive escalations based on no significant infusional toxicity or GVHD in the recipients

SUMMARY:
The purpose of the study is to determine if the use of activated T cells can effectively treat relapsed disease following allogeneic hematopoietic cell transplantation without causing GVHD.

ELIGIBILITY:
Inclusion Criteria:- Evidence of recurrent or persistent hematologic malignancy following HLA matched allogeneic hematopoietic cell transplant

* eligible for DLI
* no evidence of GVHD
* stable immunosuppressive regimen
* adequate renal and liver function Exclusion Criteria:- CML patients who have not received DLI, active infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To determine the feasibility of expanding allogeneic cytokine induced killer cells suitable for clinical application using a continuous perfusion culture system. | 21 to 28days before infusion
To determine the infusional toxicity of ex vivo expanded allogeneic CIK cells in patients with recurrent or refractory disease following allogeneic hematopoietic cell transplantation. | day of infusion up to 24 hours after infusion
To determine the incidence of Graft-versus-Host Disease (GVHD) following infusion of allogeneic CIK cells. | first 100 days after infusion
To determine the maximum tolerated dose (MTD) of expanded CIK cells for infusion. | day plus 100 after infusion

SECONDARY OUTCOMES:
o determine the incidence of disease response following treatment with allogeneic CIK cells. | one year
To assess donor-specific chimerism before and after treatment with allogeneic CIK cells. | 3 months
To optimize the ex vivo expansion of CIK cells using a continuous perfusion culture system. | 21-28 days

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Negrin, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States